CLINICAL TRIAL: NCT01240993
Title: Fostering Mothers' Emotionally-Responsive Parenting
Brief Title: Trial of Mentalization-Based Therapy for Substance Using Mothers of Infants and Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0407026890-C
Record Dates: First submitted 2010-11-05; First posted 2010-11-15 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Parenting Capacities of Substance Abusing Mothers
Keywords: parenting intervention; mother-child relations; substance abuse; attachment; child development
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parent Education (Active Comparator): PE was developed to represent parent education and support that is typically available to mothers with substance use problems who are at high risk for neglecting their young children. Mothers enrolled in PEP will meet weekly for one hour with a PE counselor who will provide assistance in solving problems related to family basic needs (e.g., health care, child care, housing and education). The PE counselor will also provide a choice of pamphlets on age-related parenting topics each week from a series of pamphlets designed specifically for this study.
  Interventions: Behavioral: Parent Education
- Mothers and Toddlers Program (Experimental): This intervention is an introductory, short-term, supportive, psychodynamic therapy for substance using mothers of young children that emphasizes the development of the capacity for mentalizing. Mothers meet with an individual, MBT-trained psychodynamically-oriented therapist for 12 sessions. The intervention is conducted a clinic where mothers are enrolled in treatment for their substance abuse.
  Interventions: Behavioral: Mothers and Toddlers Program

INTERVENTIONS:
Behavioral: Mothers and Toddlers Program — This intervention is a short-term attachment-based parenting therapy for substance using mothers of young children that emphasizes the development of the capacity for mentalizing.
  Arms: Mothers and Toddlers Program
Behavioral: Parent Education — PE was developed to represent parent education and support that is typically available to mothers with substance use problems who are at high risk for neglecting their young children. Mothers enrolled in PEP will meet weekly for one hour with a PE counselor who will provide assistance in solving problems related to family basic needs and a choice of pamphlets on age-related parenting topics.
  Arms: Parent Education

SUMMARY:
A formal randomized efficacy trial testing the Mothers and Toddlers' program, an attachment-based parenting intervention for mothers enrolled in addiction treatment and caring for young children.

DETAILED DESCRIPTION:
Five years ago the investigators were funded to develop the Mothers and Toddlers Program (MTP; R01 DA17294 / Project Period: 8/20/04 - 12/31/09). MTP is the first parenting intervention developed for substance abusing mothers based on the attachment theory. It is also the only parenting intervention for substance abusing mothers that has led to improvement in maternal caregiving sensitivity and responsiveness to infant and toddler distress in observed lab-based interactions. The investigators now have all the research materials to conduct a Stage II randomized clinical trial including a treatment manual, treatment fidelity scales therapist training program and outcome measures. In this Stage II formal efficacy trial, the investigators (1) Introduce new measures of dyadic adjustment and child attachment, (2) Add an 18 week follow up period to test for sustained treatment effects, (3) Measure major constructs (reflective functioning, representations, dyadic adjustment, and child attachment) when they are expected to change, (4) Examine temporal mechanisms of change proposed in the MTP treatment model (5) Determine whether improvements in dyadic adjustment reduces incidence of relapse, (6) Broaden the MTP therapist pool by training four new therapists and (7) Broaden the coding pool by training 3 additional coders per measure. One hundred and fifty mothers caring for children ages 12 to 60 months of age will be recruited from outpatient substance abuse treatment services at the APT Foundation into the intention-to-treat sample and will be randomized to 12 weeks of MTP vs. PEP and followed for 33 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All mothers ages 21 to 45 years, who are enrolled in treatment at one of the five APT Foundation clinics and caring for a biological child between 12 and 60 months of age will be eligible to participate.

Exclusion Criteria:

* Severe mental health problems (e.g., suicidal, homicidal, psychosis, thought disorder)
* Severe cognitive impairment
* Inability to speak English
* Target child with serious illness or significant developmental delay (e.g., cognitive, language, or motor).

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2010-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Parent Development Interview coded for maternal reflective functioning | Change at week 12 (post-treatment) from baseline
  The Parent Development Interview (PDI; Slade, Aber, Berger, Bresgi, & Kaplan, 2002) was used to measure maternal capacity to mentalize about her own and her child's behavior. The PDI is a 1 hour semi-structured interview designed to elicit the mother's narrative about commonly occurring, emotionally-challenging aspects of parenting. A rating of 1 indicates a absence of recognition of mental states. A rating of 3 indicates a limited capacity to acknowledge mental states. A rating of 5 indicates the presence of a rudimentary capacity for reflective functioning.
Parent Development Interview coded for maternal reflective functioning | Change at week 33 (follow up) from baseline
  The Parent Development Interview (PDI; Slade, Aber, Berger, Bresgi, & Kaplan, 2002) was used to measure maternal capacity to mentalize about her own and her child's behavior. The PDI is a 1 hour semi-structured interview designed to elicit the mother's narrative about commonly occurring, emotionally-challenging aspects of parenting. A rating of 1 indicates a absence of recognition of mental states. A rating of 3 indicates a limited capacity to acknowledge mental states. A rating of 5 indicates the presence of a rudimentary capacity for reflective functioning.

SECONDARY OUTCOMES:
Working Model of the Child Interview (coded for representation quality) | Change at week 12 (post-treatment) from baseline
  The Working Model of the Child Interview (WMCI; Zeanah & Benoit, 1993) is a 1.5 hour interview used to elicit a narrative description of the mother's perceptions of her child and their relationship. The rater was trained by the to reliably code 6e qualitative subscales Openness, Richness, Coherence, Caregiving Sensitivity and Acceptance and Involvement. On the mean of six subscales, a score of three is considered to represent average representational quality, scores of 1 and 2 are considered to represent clinical risk and scores of 4 and 5 are considered to represent optimal quality.
Working Model of the Child Interview (coded for representation quality) | Change at week 33 (follow up) from baseline
  The Working Model of the Child Interview (WMCI; Zeanah & Benoit, 1993) is a 1.5 hour interview used to elicit a narrative description of the mother's perceptions of her child and their relationship. The rater was trained by the to reliably code 6e qualitative subscales Openness, Richness, Coherence, Caregiving Sensitivity and Acceptance and Involvement. On the mean of six subscales, a score of three is considered to represent average representational quality, scores of 1 and 2 are considered to represent clinical risk and scores of 4 and 5 are considered to represent optimal quality.
NCAST Teaching Scales (Maternal Behavior) | Change at week 12 (post-treatment) from baseline
  The NCAST Teaching Scale (Barnard & Eyres, 1979) is a standardized, 73 item tool used to observe and rate quality of interactions with children birth to 36 months. Mothers choose a task to teach the child in a 5 minute teaching session. Maternal behavior is coded on 4 dimensions: Sensitivity to Cues, Response to Distress, Social-Emotional Growth Fostering, & Cognitive Growth Fostering. The Total Caregiver Score is the sum of the 4 subscale scores. The Total Caregiver Contingency Score is the sum of 20 items from the 4 subscales that involve the caregiver's contingent response to child cues.
NCAST Teaching Scales (Maternal Behavior) | Change at week 33 (follow up) from baseline
  The NCAST Teaching Scale (Barnard & Eyres, 1979) is a standardized, 73 item tool used to observe and rate quality of interactions with children birth to 36 months. Mothers choose a task to teach the child in a 5 minute teaching session. Maternal behavior is coded on 4 dimensions: Sensitivity to Cues, Response to Distress, Social-Emotional Growth Fostering, & Cognitive Growth Fostering. The Total Caregiver Score is the sum of the 4 subscale scores. The Total Caregiver Contingency Score is the sum of 20 items from the 4 subscales that involve the caregiver's contingent response to child cues.
NCAST Teaching Scales (Child Behavior) | Change at week 12 (post-treatment) from baseline
  Child behavior with the mother was assessed using the Clarity of Cues and the Responsiveness to Caregiver Subscales from the NCAST Teaching Scales. The Child Total Score is the sum of the 2 scales. The Child Contingency Score is the sum of 12 contingent items from the 2 scales.
NCAST Teaching Scales (Child Behavior) | Change at week 33 (follow up) from baseline
  Child behavior with the mother was assessed using the Clarity of Cues and the Responsiveness to Caregiver Subscales from the NCAST Teaching Scales. The Child Total Score is the sum of the 2 scales. The Child Contingency Score is the sum of 12 contingent items from the 2 scales.
Child Attachment Status | Change at week 12 (post-treatment) from baseline
  We will use the standard 8-episode protocol Strange Situation protocol. Each child will receive a classification of secure, insecure or disorganized for each time point.
Beck Depression Inventory | Change at week 12 (post-treatment) from baseline
  The Beck Depression Inventory (BDI; Beck, Steer, & Brown, 1996) was used to assess maternal symptoms of depression. The BDI is a widely used 21-item questionnaire rated on a 4-point scale and yields a total score ranging from 0 to 63: scores between 13 and 19 indicate mild depression; scores between 20 and 28 indicate moderate levels of depression, and scores between 29 and 63 indicate severe levels of depression (Beck et al., 1996).
Beck Depression Inventory | Change at week 33 (follow up) from baseline
  The Beck Depression Inventory (BDI; Beck, Steer, & Brown, 1996) was used to assess maternal symptoms of depression. The BDI is a widely used 21-item questionnaire rated on a 4-point scale and yields a total score ranging from 0 to 63: scores between 13 and 19 indicate mild depression; scores between 20 and 28 indicate moderate levels of depression, and scores between 29 and 63 indicate severe levels of depression (Beck et al., 1996).
Brief Symptom Inventory | Change at week 33 (follow up) from baseline
  The Brief Symptom Inventory (BSI; Derogatis, 1993) was used to assess maternal global psychiatric distress. The BSI is a standardized, widely used, 53-item, 5-point, self-report measure of psychopathology. The composite Global Severity Index (GSI) measures current overall symptomatology across multiple domains and has demonstrated good reliability and validity (Derogatis, 1993). T scores above 60 on the GSI indicate risk for a clinical disorder.
Curiosity Box Paradigm | Change at week 12 (post-treatment) from baseline
  . We will use the Curiosity Box Paradigm (Mayes et al., 1993) to assess dyadic adjustment under circumstances of mild uncertainty (i.e., during the child's exploration of unfamiliar toys/objects). Children will explore a box of 9 novel toys or objects (that they are unlikely to have seen before) after an initial 5 minute warm up period with one box of 9 familiar toys. Maternal, child and dyadic behavior will be assessed with the Coding Interaction Behavior Scales (Feldman, 1998).
Curiosity Box Paradigm | Change at week 33 (follow up) from baseline
  . We will use the Curiosity Box Paradigm (Mayes et al., 1993) to assess dyadic adjustment under circumstances of mild uncertainty (i.e., during the child's exploration of unfamiliar toys/objects). Children will explore a box of 9 novel toys or objects (that they are unlikely to have seen before) after an initial 5 minute warm up period with one box of 9 familiar toys. Maternal, child and dyadic behavior will be assessed with the Coding Interaction Behavior Scales (Feldman, 1998).

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E. Suchman, Ph.D., Principal Investigator — Yale University School of Medicine, Department of Psychiatry
Locations (2):
- United States (2):
  - The Moms 'n' Kids Program at the APT Foundation, New Haven, Connecticut
  - Yale Psychosocial Substance Abuse Research Unit, West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suchman NE, DeCoste C, Castiglioni N, McMahon TJ, Rounsaville B, Mayes L. The Mothers and Toddlers Program, an attachment-based parenting intervention for substance using women: post-treatment results from a randomized clinical pilot. Attach Hum Dev. 2010 Sep;12(5):483-504. doi: 10.1080/14616734.2010.501983. PMID 20730641
- [Background] Suchman NE, DeCoste C, Leigh D, Borelli J. Reflective functioning in mothers with drug use disorders: implications for dyadic interactions with infants and toddlers. Attach Hum Dev. 2010 Nov;12(6):567-85. doi: 10.1080/14616734.2010.501988. PMID 20931415
- [Background] Suchman NE, Decoste C, McMahon TJ, Rounsaville B, Mayes L. THE MOTHERS AND TODDLERS PROGRAM, AN ATTACHMENT-BASED PARENTING INTERVENTION FOR SUBSTANCE-USING WOMEN: RESULTS AT 6-WEEK FOLLOW-UP IN A RANDOMIZED CLINICAL PILOT. Infant Ment Health J. 2011 Jul;32(4):427-449. doi: 10.1002/imhj.20303. Epub 2011 Jun 14. PMID 22685361
- [Background] Suchman N, Decoste C, Castiglioni N, Legow N, Mayes L. THE MOTHERS AND TODDLERS PROGRAM: Preliminary Findings From an Attachment-Based Parenting Intervention for Substance-Abusing Mothers. Psychoanal Psychol. 2008 Jul 1;25(3):499-517. doi: 10.1037/0736-9735.25.3.499. PMID 20057923
- [Background] Suchman NE, Decoste C, Rosenberger P, McMahon TJ. ATTACHMENT-BASED INTERVENTION FOR SUBSTANCE-USING MOTHERS: A PRELIMINARY TEST OF THE PROPOSED MECHANISMS OF CHANGE. Infant Ment Health J. 2012 Jul 1;33(4):360-371. doi: 10.1002/imhj.21311. Epub 2012 Apr 24. PMID 23024442
- [Background] Borelli JL, West JL, Decoste C, Suchman NE. EMOTIONALLY AVOIDANT LANGUAGE IN THE PARENTING INTERVIEWS OF SUBSTANCE-DEPENDENT MOTHERS: ASSOCIATIONS WITH REFLECTIVE FUNCTIONING, RECENT SUBSTANCE USE, AND PARENTING BEHAVIOR. Infant Ment Health J. 2012;33(5):506-519. doi: 10.1002/imhj.21340. Epub 2012 May 22. PMID 23049148
- [Result] Suchman NE, DeCoste CL, McMahon TJ, Dalton R, Mayes LC, Borelli J. Mothering From the Inside Out: Results of a second randomized clinical trial testing a mentalization-based intervention for mothers in addiction treatment. Dev Psychopathol. 2017 May;29(2):617-636. doi: 10.1017/S0954579417000220. PMID 28401850
- [Result] Suchman NE. Mothering from the Inside Out: A mentalization-based therapy for mothers in treatment for drug addiction. Int J Birth Parent Educ. 2016 Jul;3(4):19-24. PMID 27840685
- [Result] Suchman NE, DeCoste C, Borelli JL, McMahon TJ. Does improvement in maternal attachment representations predict greater maternal sensitivity, child attachment security and lower rates of relapse to substance use? A second test of Mothering from the Inside Out treatment mechanisms. J Subst Abuse Treat. 2018 Feb;85:21-30. doi: 10.1016/j.jsat.2017.11.006. Epub 2017 Nov 21. PMID 29291768